CLINICAL TRIAL: NCT05402891
Title: The Chemopreventive Effect of Lithium on Adenoma Development in Patients With Familial Adenomatous Polyposis (FAP); a Pilot Study
Brief Title: The CHAMP-study: The CHemopreventive Effect of Lithium in Familial AdenoMatous Polyposis
Acronym: Lithium in FAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL80308.018.22
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Familial Adenomatous Polyposis; Chemopreventive therapy; Adenoma development; Lithium carbonate
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Lithium Carbonate

STUDY DESIGN:
Intervention Model Description: A prospective phase II, single arm pilot trial, with a duration of 18 months. The drug will be administered between month 6 and 12. All patients will be treated with Lithium with an oral dose of 300mg a day for six months, achieving a therapeutic serum level between 0.2-0.4 mmol/L. The duration of this study will be 18 months, and patients will undergo four colonoscopies in total (at t=0, t=6, t=12, t=18). During each colonoscopy biopsies from normal intestinal mucosa will be collected to determine stem cell dynamics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study population (Experimental): Every patient will receive treatment: Lithiumcarbonate 300mg daily in oral tablet for six months. There will no control group included since patient represent their own control in the nontreatment-phase.
  Interventions: Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate — Patients will be administered lithiumcarbonate by an oral tablet of 300mg once a day for a duration of 6 months. Starting dose is 200mg for the first 5 days, dosage will be then increased to 300mg. To limit adverse events and side-effects, the lowest effective dose will be administered. The target serum level of lithium is 0.20 - 0.40 mmol/L and this will be maintained by regular lithium level testing.

SUMMARY:
Rationale: Familial adenomatous polyposis (FAP) syndrome is characterized by the development of numerous colorectal polyps. If left untreated, these patients have a chance of nearly 100% of developing colorectal cancer (CRC) at a young age. Therefore, guidelines recommend a prophylactic colectomy during early adulthood. Even after colectomy, most patients will develop adenomas in the retained rectum or ileoanal pouch requiring further endoscopic surveillance. In a recent study in mouse models, a chemopreventive effect of Lithium was observed on the spread of Apc mutated cells within the crypts of normal intestinal mucosa, suggesting polyp formation can be prevented. Lithium is used to treat patients with bipolar disorders but has never been investigated in patients with FAP aiming to reduce polyp burden. We hypothesize that Lithium could reduce the spread of APC mutated cells within the crypt of normal intestinal mucosa potentially reducing polyp burden in patients with FAP.

Objective: The aim of this study is to investigate the effect of low-dose Lithium on stem cell dynamics, the number and size of polyps and, to assess safety outcomes of this drug in FAP patients.

Study design: A prospective phase II, single arm pilot trial, with a duration of 18 months. The drug will be administered between month 6 and 12.

Study population: Twelve patients with FAP between the age of 18 and 35 not having undergone a colectomy (yet), having a genetically confirmed APC mutation and a family history with a classical FAP phenotype.

Intervention: All patients will be treated with Lithium with an oral dose of 300mg a day for six months, achieving a therapeutic serum level between 0.2-0.4 mmol/L.

Main study parameters/endpoints: The main outcome parameter is the effect of Lithium on the spread of APC mutant cells within intestinal crypts over time by using an APC specific marker NOTUM (a significance reduce of fixed crypts and reduction of fixed clone size of 50%).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: A physical examination and an endoscopy with biopsies will be performed at baseline and every six months (four in total). Laboratory testing will be done at baseline and every two months during Lithium treatment. Patients will be interviewed by phone and Lithium side effect questionnaires will be obtained at baseline and during Lithium treatment. Lithium serum levels will be measured at day 12 and 22 after start of the study drug (at month 6). When the therapeutic range has been achieved, serum level testing will be done every month. Most relevant side-effects that could potential occur include polyuria, hyperparathyroidism and hypothyroidism. Most side effects are dose-dependent and will be regularly monitored. Patients with FAP could potentially benefit from a chemopreventive therapy such as Lithium to postpone or even avoid invasive types of surgery.

DETAILED DESCRIPTION:
For this study, monitoring was requested from Clinical Monitoring Center (CMC). After approval by the METC, a monitoring intake visit will be scheduled to set up a monitoring plan.

In this study, no randomisation will take place, every participant is given the same treatment.

All crypt analysis data and adenoma counts will be scored blindly.

Patients will be recruited from the large cohort of FAP patients at the hereditary GI Cancer clinic at the Amsterdam UMC. Prior to their routine surveillance colonoscopy, patients will be invited to participate by a member of the study team. In total 12 patients will be included in this trial.

Adenomatous tissue collected endoscopically, as part of routine care, will be stored according to regulations of the department of pathology in the AMC. Normal intestinal mucosa collected endoscopically, as part of study material to assess NOTUM distribution size e.g., will be analysed in the Center for Experimental and Molecular Medicine (CEMM). Source documents and CRFs will be stored by the project leader for 15 years after closure of the trial. Collected samples will be stored for 5 years. In case of informed consent is reached for participation in a biobank, samples will be stored for 15 years. Data of the subjects will be coded in order of participation. The code and the data are stored in different locations. The code can only be seen by the investigators. Qualified authorities can get insight in the code and data, but only when accompanied by the investigators. Informed consent forms are kept in separate files, to ensure the data security. The handling of personal data will comply with the Dutch Personal Data Protection Act.

Since this study is not yet been performed in humans with FAP, this study will be a pilot study. We believe a number of 12 patients is sufficient for the explorative purpose of this study. By performing a paired analysis, the effect of variation between individuals will be reduced, and we expect sufficient power to draw significant results. To detect a reduction of 50% (power stat. 80%, p=0.05) in fitness of APC-mutant cells, we need to analyse sizes of APC mutant clones within 11 partially populated crypts. To ensure sufficient material we need 840 crypts per patient per time point. A typical biopsy yields 100-250 crypts, therefore we will perform 12 biopsies in total (2 biopsies per segment, 6 segments) per patient per time point. In that way, sufficient data will be obtained to confirm or refute the study hypothesis.

Subjects who withdraw from the trial after start of Lithiumcarbonate will not be replaced.

To describe the study population, baseline characteristics and changes in outcome parameters during follow-up, descriptive statistics will be used in this study. SPSS for Windows software (Chicago, IL, USA) version 26.0 will be used for these analyses. If other statistical analysis will be used, this will be mentioned in the study paper.

Primary analysis for the primary outcome parameter will be done by analyzing the data using two-sided student's t-test. will be performed. The limit for the statistical significance will be established at p < 0.05 with a confidence interval of 95%.

Descriptive statistics will be used to describe the changes in outcome measures during follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria for inclusion in the study:

* Age between 18 and 35 years;
* Confirmed APC germline mutation and one of the following:

  * Minimum of 100 colorectal adenomas
  * Minimum of 50 colorectal adenomas and a positive family history of a classical FAP phenotype (>100 colorectal adenomas);
* Intact colon;
* Participant is willing and able to give informed consent for participation.

Exclusion Criteria:

Patients that meets any of the following criteria will be excluded from participation in this study:

* Participation in any other clinical intervention study; observational trials accepted;
* Lithium use prior to participation of the study;
* Pregnancy, breast-feeding or no use of anticonception;
* No normal intestinal mucosa left for normal tissue biopsy;
* Indication for colectomy within 2 years;
* Known renal impairment, defined as GFR < 60 ml/min;
* Known severe cardiac disorder;
* Known severe brain injury;
* Hypothyroidism;
* Hyponatremia, defined as Na < 130mmol/L;
* Positive family history of Brugada syndrome
* Co-medication known for interacting with lithium
* Regular NSAID use (defined as more than twice a week for 4 consecutive weeks) within 3 months prior to baseline;
* Use of immunosuppressive or anti-inflammatory drugs within 3 months prior to baseline;
* Use of any other FAP directed drug therapy within 3 months prior to baseline (use of any alternative supplements e.g. turmeric or fish-oil must be noted in questionnaire).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in clone size distribution positive for NOTUM. | Month 0, Month 6, Month 12, Month 18
  For each patient crypts will be retrieved form normal tissue biopsies through colonoscopy. APC mutant stem cell dynamics will be determined by tracing the spread of the APC mutant cells using specific expression of NOTUM by RNAscope (in situ hybridization). Clone sizes will be quantified as proportions of the crypt circumference positive for NOTUM (in parts of eight, 1:8 to 8:8). When a whole crypt is positive for NOTUM (8:8), this crypt is fixed (crypt fixation) (12). This will result in an average clone size distribution for each patient per time point, as well as the proportion of fixed crypts. By analyzing the differences in clone size distribution before, during and after Lithiumcarbonate treatment we aim to observe a relative reduction in average clone size of 50% during the lithiumcarbonate treatment, as well as a reduction in crypt fixation of 50%.

SECONDARY OUTCOMES:
Change in number and size of polyps (defined as polyp burden) | Month 0, Month 6, Month 12, Month 18
  A full colonoscopy will be performed to assess polyp burden and take biopsies. During colonoscopy, BBPS should be 2 for each segment and cecal intubation achieved. Adenoma burden will be assessed by estimating the number and size (estimated using a biopsy forceps) of adenomas in each of the 6 colorectal segments: cecum, ascending colon, transverse colon, descending colon, sigmoid and rectum (including retroflexion). Size of polyps is divided into groups of 1-2mm, 3-5mm, 6-10mm, >10mm. The number per size is added up to outcome measure 'polypburden'. Standard white light endoscopy (WLE) will be used; NBI is used at the discretion of the endoscopist. Video recordings will be made for all colonoscopies (only using WLE). All four videos of each participant will be reviewed by two separate independent expert endoscopists in a random order, assessing the adenoma burden.
Patient reported side effects of Lithiumcarbonate using a Lithium side effect questionnaire | Month 0, Month 6 (day 22), Month 9
Safety outcomes by analysing reported adverse events, physical examination and laboratory findings. | Physical examination (including vital signs) at baseline and every six months (at time of endoscopy). Interviewing: month 0, month 3, month 6, month 7, month 9, month 11, month 12, month 15, month 18, month 19. Laboratory testing will be done at baseline

OTHER OUTCOMES:
Number of cups of coffee per day (decaffeinated coffee not included) | month 0, month 3, month 6, month 7, month 9, month 11, month 12, month 15, month 18
  By using a diet diary
Turmeric use (gram per day) | month 0, month 3, month 6, month 7, month 9, month 11, month 12, month 15, month 18
  By using a diet diary
Number of fish oil capsules per day (amount of eicosapentaenoic acid in terms of mg) | month 0, month 3, month 6, month 7, month 9, month 11, month 12, month 15, month 18
  By using a diet diary
History of smoking, if yes number of pack years | Month 0

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Neerven SM, de Groot NE, Nijman LE, Scicluna BP, van Driel MS, Lecca MC, Warmerdam DO, Kakkar V, Moreno LF, Vieira Braga FA, Sanches DR, Ramesh P, Ten Hoorn S, Aelvoet AS, van Boxel MF, Koens L, Krawczyk PM, Koster J, Dekker E, Medema JP, Winton DJ, Bijlsma MF, Morrissey E, Leveille N, Vermeulen L. Apc-mutant cells act as supercompetitors in intestinal tumour initiation. Nature. 2021 Jun;594(7863):436-441. doi: 10.1038/s41586-021-03558-4. Epub 2021 Jun 2. PMID 34079128
- [Derived] Linssen JDG, van Neerven SM, Aelvoet AS, Elbers CC, Vermeulen L, Dekker E. The CHAMP-study: the CHemopreventive effect of lithium in familial AdenoMatous Polyposis; study protocol of a phase II trial. BMC Gastroenterol. 2022 Aug 12;22(1):383. doi: 10.1186/s12876-022-02442-3. PMID 35962368

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT05402891/Prot_SAP_000.pdf